CLINICAL TRIAL: NCT00775073
Title: Antiangiogenic Treatment of Advanced or Metastatic Hepatocellular Cancer (HCC) - An Open Label, Stratified, Single-arm Phase II Study of Bevacizumab and RAD001
Brief Title: Antiangiogenic Treatment of Hepatocellular Cancer With Bevacizumab and RAD001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gerhard Treiber (Individual)
Collaborators: Crolll Gmbh (Other); Estimate, GmbH (Industry); Janssen Diagnostics, LLC (Industry)
Responsible Party: Sponsor-Investigator, Gerhard Treiber, Prof. Dr. med., Treiber, Gerhard
Organization: Treiber, Gerhard (Individual)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001C24100
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Liver cancer; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Everolimus; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Bevacizumab (Avastin) & Everolimus (RAD001)
  Interventions: Drug: Everolimus, Bevacizumab

INTERVENTIONS:
Drug: Everolimus, Bevacizumab — Everolimus 5 mg tablet per day orally. Bevazicumab 5 mg per kg intravenous every 2 weeks.
  Other Names: RAD001; Avastin

SUMMARY:
This is a prospective open label clinical trial in patients with advanced or metastatic liver cancer to assess the clinical and biological activity of RAD001 (Everolimus) in conjunction with Bevazicumab (Avastin). Approximately 36 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients with non-resectable locally advanced or metastatic hepatocellular cancer BCLC stage B and C. BCLC stage A can occasionally be included provided that other treatment options are unavailable
* Measurable disease: At least one measurable lesion (longest diameter ≥20 mm on conventional CT or MRI scan; ≥ 10 mm on spiral CT) according to RECIST criteria that has not been previously locally treated by irradiation, surgery, ethanol injection, radiofrequency ablation or transarterial chemoembolisation
* Confirmation of HCC disease by histology (preceding liver resection or fine needle biopsy within the last 12 months);
* Liver Function: Child A and B
* Tumor extent: CLIP Score ≤ 3
* ECOG Performance Status 0-2 (=Karnofsky-Index ≥ 60%)

Exclusion Criteria:

* Patient had received any prior systemic treatment (possible exception: sorafenib for a maximum of 3 months, last dose received at least 28 days before study inclusion)
* Patient had a major surgery, local ablative treatments (RFA, PEI), or transarterial chemoembolisation therapy within 4 weeks prior to randomisation
* Presence of a secondary malignancy either at the time of screening or in the past 5 years: An exception from this rule can be made in patients that were treated in curative intention within the last 3 years and are without any evidence of recurrence of this malignancy.
* History or presence of central nervous system (CNS) disease (i.e., primary brain tumor, malignant seizures, CNS metastases or carcinomatous meningitis) or other mental illness.
* Clinically serious infections or uncontrolled infection (including HIV infection), increased risk for acquisition of opportunistic infections
* Chronic treatment with systemic steroids or another immunosuppressive agent
* Inadequate organ functions, characterised by: cholestasis with elevated levels of bilirubin and/or alkaline phosphatase > 3x UNL (can be improved by biliary drainage if necessary) and/or elevated transaminases (ALAT/ASAT) ≥ 5 x UNL, hypoalbuminemia < 2.5 g/dl, renal impairment (serum creatinine < 1.5 x UNL ), inadequate Hematology: Platelets < 75.000, ANC < 1500, hemoglobin < 9.0 mg/dl, inadequate coagulation status, namely INR > 2 or Quick < 50%, aPTT >50 sec in the absence of any drugs interfering with coagulation such as warfarin, phenprocoumon, NMH or UFH. Fasting serum cholesterol ≤300 mg/dL OR 7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN, patients with severe refractory therapy-resistant hyperlipidemia
* Women who are pregnant or breast feeding, intended pregnancy, or women unable to conceive and unwilling to practice an effective method of birth control
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of RAD001 and cannot be controlled by adequate medical treatment (e.g. uncontrolled nausea, vomiting, diarrhoea which might result in malabsorption, any known malabsorption syndrome, bowel obstruction, or inability to swallow the capsules/tablets)

Exclusion Criteria derived from special situations:

* Mixed tumors of HCC with cholangiocarcinoma or fibrolamellar HCC type
* Patients with complications of liver cirrhosis such as recent spontaneous bacterial infection of ascites, hepatic encephalopathy > grade 2 during the last 2 weeks and not adequately controlled or hepatorenal syndrome not responding to conservative treatment within 2 weeks
* Patients with any active gastrointestinal bleeding during the last 2 weeks
* Patients without screening EGD during the last 2 weeks
* Patients with nonbleeding gastroesophageal varices grade I° with red coloured signs or grade ≥ II° on EGD that do not undergo prophylactic ligation or sclerosing treatment at least one week before the first dose of study medication is taken.
* Patients with unhealed gastrointestinal ulcerations or wounds
* Patients with a history of one of the following: bowel perforation, colon diverticulitis
* Any relevant findings on screening colonoscopy
* History of any thromboembolic events (except for portal vein infiltration and/or thrombosis)
* Allergic reactions or intolerance to previous drug exposure to RAD001 or bevacizumab; having received any of the study medications within the last 3 years before randomisation
* Allergy or intolerance against CHO-cell products or other recombinant human or humanised antibodies
* Patients with an increased risk for the development of lymphoma or other malignant diseases, especially concerning the skin
* Patients with rare hereditary disorders like galactose intolerance, lactase deficiency or glucose-galactose malabsorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-10; Primary Completion 2011-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Time to Progression | 24 and 48 weeks

SECONDARY OUTCOMES:
Overall Survival | 24 and 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Treiber, PD Dr., Principal Investigator — Zollernalbklinikum Balingen
Locations (10):
- Germany (10):
  - Medizinische Klinik 1 University of Erlangen, Erlangen, Bavaria
  - Zollernalbklinikum, Balingen
  - Charité, Campus Virchow Klinikum, Medizinische Klinik mit Schwerpunkt Hepatologie und Gastroenterologie, Berlin
  - Universitaetsklinikum Bonn, Medizinische Klinik und Poliklinik I, Bonn
  - Klinikum der J.-W.-Goethe-Universitaet, Medizinische Klinik I, Frankfurt
  - Medizinische Universitaetsklinik Freiburg, Innere Medizin II, Freiburg im Breisgau
  - Martin-Luther-Universitaet Halle-Wittenberg, Universitaetsklinik und Poliklinik für Innere Medizin I, Halle
  - Medizinische Hochschule Hannover, Zentrum Innere Medizin, Hanover
  - Universitätsklinikum des Saarlandes Klinik für Innere medizin II, Homburg/Saar
  - Medizinische Fakultaet der Otto-von-Guericke-Universitaet, Klinik für Gastroenterologie, Hepatologie und Infektiologie, Magdeburg

REFERENCES:
- [Derived] Treiber G. mTOR inhibitors for hepatocellular cancer: a forward-moving target. Expert Rev Anticancer Ther. 2009 Feb;9(2):247-61. doi: 10.1586/14737140.9.2.247. PMID 19192962